CLINICAL TRIAL: NCT05917028
Title: A Single Arm, Single Center, Open Label , Pilot Clinical Study to Evaluate the Efficacy and Safety of Transcatheter Arterial Micro Embolization (TAME) Using Nexsphere F in Patients With Knee Degenerative Osteoarthritis
Brief Title: Transcatheter Arterial Micro-Embolization (TAME) Using Nexsphere-F in Patients With Knee Degenerative Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Next Biomedical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NS-F TAME001
Record Dates: First submitted 2023-06-12; First posted 2023-06-23 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Transcatheter Arterial Micro-Embolization (Experimental): If abnormal blood vessels related to pain are identified by angiography, selective embolization is performed using Nexsphere-F.
  Interventions: Device: Transcatheter Arterial Micro-Embolization

INTERVENTIONS:
Device: Transcatheter Arterial Micro-Embolization — Participants will undergo TAME with Nexsphere-F.

SUMMARY:
Among knee degenerative osteoarthritis patients aged 50 or older, it will prove the therapeutic effect and safety of Nexsphere-F embolization for patients who need additional treatment because pain is not controlled even if conventional treatments are taken.

DETAILED DESCRIPTION:
This clinical trial is a single arm, single center, open label, and pilot clinical trial to prove the performance and safety of Nexsphere-F in patients over the age of 50 who need additional treatment because pain is not controlled even after conventional treatments are taken.

Since consent cannot be obtained during surgery from a subject who meets the inclusion and exclusion criteria, a written consent is obtained in advance between four weeks before the procedure and the day. As one of the usual orthopedic evaluations, baseline MRI will be performed and WORMS will be evaluated. In addition, the WOMAC score and the VAS score will be measured before the procedure and used as a baseline for evaluation variables. Since it is a pilot study to evaluate the validity, all subjects will undergo a Transcatheter Arterial Micro-Embolization (TAME).

ELIGIBILITY:
Inclusion Criteria:

* Those who fall under Kellgren-Lawrence grade 2 to 3 according to the criteria in accordance with ACR guidelines and X-ray findings used within 12 months
* VAS score exceeding 50mm
* An adult male and female over 50 years of age
* Preservative therapy Glucosamine chondroitin sulfate/physiological therapy and rehabilitation exercises, and joint injections of hyaluronic acid for more than 12 weeks
* A person who agrees to maintain existing medication treatments during the clinical trial period but does not receive additional medication or new conservative treatments for knee osteoarthritis pain management.

Exclusion Criteria:

* A locally infected patient
* A person whose life expectancy is less than six months
* A person with symptoms of lower extremities that are considered secondary to atherosclerosis or arterial vascular disease (ex: claudication ischemic rest pain)
* A person diagnosed with rheumatism or infectious arthritis
* A person who has undergone knee arthroplasty
* A person who has not had knee microfracture surgery for more than 10 years
* INR 2.5 or less than 30,000 platelets
* Anaphylaxis-causing iodine allergy
* Patients with renal dysfunction or impaired renal function who have been diagnosed with less than 45 GFR (eGFR) within the last 60 days
* Those who have a taboo on MR videos
* Pregnant women
* Other cases where it is deemed inappropriate to participate in this clinical trial at the discretion of the researcher

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-10-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Rate of WOMAC Score Reduction | 1 day, 14 days, 1 month, 3 months, 6 months
  The rate of change of WOMAC Score before and after application of medical devices for clinical trials. The definition of clinical success is a reduction of more than 50% of baseline scores (WOMAC and VAS) in six-month observations after at least one knee vascular embolization without additional combination treatment.
Rate of VAS Score (patient pain intensity) Reduction | 1 day, 14 days, 1 month, 3 months, 6 months
  The rate of change of VAS Score before and after application of medical devices for clinical trials. The definition of clinical success is a reduction of more than 50% of baseline scores (WOMAC and VAS) in six-month observations after at least one knee vascular embolization without additional combination treatment.

SECONDARY OUTCOMES:
Rate of change in WORMS (Whole-Organ Magnetic Resonance Imaging Score) | 1 month
  The rate of change of WORMS before and after application of medical devices for clinical trials. MRI images of cartilage, marrow abnormality, bone cysts, bone attrition, ostephytes, menisci, ligaments, and synovitis are scored and recorded.
The rate of reduction of medication | 6 months
  The rate of change of medication before and after application of medical devices for clinical trials.
The rate of discontinuation of combination treatment | 6 months
  The rate of change of combination treatment before and after application of medical devices for clinical trials.

OTHER OUTCOMES:
Number of participants with abnormal cases during follow-up (AVN, skin necrosis, dermal toxicity, acute lower extremity ischemia) | 1 day, 14 days, 1 month, 3 months, 6 months
  Abnormal cases that occurred after the application of medical devices for clinical trials (AVN, skin necrosis, dermal toxicity, acute lower extremity ischemia)

CONTACTS AND LOCATIONS:
Overall Officials: Hyuckmin Kwon, Principal Investigator — Severance Hospital
Locations (1):
- Severance Hospital, Seoul, Seodaemun-gu, South Korea

IPD SHARING:
Plan to Share IPD: No